CLINICAL TRIAL: NCT03453047
Title: Evaluation of Preoperative and Postoperative S100β and Neuron Specific Enolase Levels in Patients Undergoing Liver Transplantation
Brief Title: S100β and Neuron Specific Enolase Levels in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Bora Dinc (Other)
Responsible Party: Sponsor-Investigator, Bora Dinc, Assistant Professor Department of Anesthesiology and Reanimation, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: LIVER
Record Dates: First submitted 2018-01-30; First posted 2018-03-05 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Liver Transplantation
Keywords: S100β; Neuron specific enolase; Liver transplantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — analyzing S100β and neuron specific enolase serum concentrations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Healthy volunteers. Liver donor groups; Course of the research: Blood samples from all groups shall be taken for S100β and NSE in preoperative period, in the operating room and after 1 and 6 months in postoperative period. Mortality and morbidity of the patients shall be recorded. Neurological damage and its effect on prognosis shall be examined within the patients who were transplanted liver with S100β and NSE. Demographic data of the patients, accompanying diseases, American Society of Anesthesia classification, etiology, Model For End-Stage Liver Disease score, Child classification, sodium, potassium, total bilirubin, alanine aminotransferase, aspartate aminotransferase, Alkaline phosphatase, International Normalized Ratio, creatinine and urea shall be recorded. Intraoperative medicine administration and fluid balance, duration of operation, graft hot ischemia and graft cold ischemia durations, initial pulmonary artery pressure, blood component transplantations shall be recorded.
  Interventions: Diagnostic Test: S100β and Neuron specific enolase (NSE)
- 2: Liver transplant groups;Course of the research Blood samples from all groups shall be taken for S100β and NSE in preoperative period, in the operating room and after 1 and 6 months in postoperative period. Mortality and morbidity of the patients shall be recorded. Neurological damage and its effect on prognosis shall be examined within the patients who were transplanted liver with S100β and NSE. Demographic data of the patients, accompanying diseases, American Society of Anesthesia classification, etiology, Model For End-Stage Liver Disease score, Child classification, sodium, potassium, total bilirubin, alanine aminotransferase, aspartate aminotransferase, Alkaline phosphatase, International Normalized Ratio, creatinine and urea shall be recorded. Intraoperative medicine administration and fluid balance, duration of operation, graft hot ischemia and graft cold ischemia durations, initial pulmonary artery pressure, blood component transplantations shall be recorded.
  Interventions: Diagnostic Test: S100β and Neuron specific enolase (NSE)

INTERVENTIONS:
Diagnostic Test: S100β and Neuron specific enolase (NSE) — S100β is 10.4 kDa protein. Synthesized with end feet processes of astrocytes in the brain S100β belongs to low molecular weight EF-hand type acidic calcium binding protein superfamily. This protein is metabolized in the kidneys and removed with urine. It is shown that S100β does not show differences due to ethnical groups or genders and is not affected by circadian rhythm. Although S100β is also found in other tissues, it is in higher concentrations in the brain so it can be used as an early indicator for brain damage.NSE is an SSS protein which exists in neurons and neuroendocrine tissues. NSE plays a role in glycolytic route in neurons as intracytoplasmic enzyme increasing serum level in case of neuron damage. Whilst S100β is the marker of astroglia dysfunction, NSE is the marker of neuronal dysfunction.

SUMMARY:
Several neurological problems which include both central nervous system and peripheral nervous system can occur as a result of acute liver failure or severe chronic liver failure. The main reason of cerebral damage in liver failure is cellular metabolic changes, long term neuro-inflammation status, activation of brain microglia, accumulation of manganese and ammonia besides acute and severe hyperammoniemia that triggers systemic inflammation. Examples of neurological complications of serious hepatocellular failure are hepatic encephalopathy, diffuse brain edema, Wilson disease, hepatic myelopathy, acquired hepatocerebral degeneration; Parkinsonism induced cirrhosis and osmatic demyelinization. Attentive neurological evaluation is of high importance in order to define seriousness level and distribution of neurologic disorders besides current treatable anomalies and potentially prescribe postoperative prognosis.

S100β is released by astrocytes in brain damage. S100β increases in the beginning of brain damage so it can be used to diagnose early stage brain damage. Neuron specific enolase (NSE) acts as intracytoplasmic enzyme and increases serum levels in neuron damage.

The aim of the study is to evaluate neurological damage and analyze its effect on prognosis by considering S100β and NSE levels in liver transplantation.

DETAILED DESCRIPTION:
Neurologic disorders that affect the liver transplantation candidates when they are on the waitlist not only significantly affect preoperative morbidity and even mortality but also present important predictive factors for post-op neurologic manifestations. Attentive neurological evaluation before transplantation plays a significant role in defining seriousness level and distribution of neurologic disorders besides current treatable anomalies and potentially prescribe postoperative prognosis. Preferred specific indexes of neurological evaluation before transplantation can vary according to centers but correct diagnosis and definitive diagnosis of some syndromes can be difficult despite using current biochemical, neurophysiologic, neuropsychological and neuroimaging diagnosis tools.

Liver transplant receivers constitute the group with the most frequent central nervous system complication (incidence: 10%-85%) amongst the organ transplantation patients. They are focal or diffuse neurologic deficits creating a significant obstacle for short and long term recovery. Neurologic deficits which can develop are cerebral edema, increase of intracranial pressure, metabolic encephalopathy, cerebrovascular complications, osmotic demyelination syndrome and opportunistic infections. Moreover, several preoperative neurologic disorders (such as dysarthria akinetic mutism, confusion and seizures) can get worse due to neurotoxic side effect of the medicines which are used for preventing graft rejection (calcineurin inhibitors).

Neurologic findings and pathophysiology of end stage liver failure cannot be understood completely. Multiple factors such as long term brain "neuroinflammation", brain microglia, activation of inflammatory cells, accumulation of manganese and ammonia, changing blood-brain barrier permeability, changed nerve conduction and inflammation of peripheric nerve system inflammation are held responsible from brain damage. Other negative direct or indirect neurologic effects are chronical malnutrition, gastrointestinal bleeding, cerebral hypoperfusion and renal dysfunction. The most commonly accepted neurological complications of serious hepatocellular insufficiency are complex syndromes of hepatic encephalopathy (HE).

S100β is 10.4 kDa (kilodalton) protein. Synthesized with end feet processes of astrocytes in the brain S100β belongs to low molecular weight EF-hand type acidic calcium binding protein superfamily. This protein is metabolized in the kidneys and removed with urine. It is shown that S100β does not show differences due to ethnical groups or genders and is not affected by circadian rhythm. Although S100β is also found in other tissues, it is in higher concentrations in the brain so it can be used as an early indicator for brain damage.

Astrocytes are the keys to homeostasis regulation in central nervous system (CNS) and release S100β after brain damage. Some studies conducted that, increased S100β levels as an early indicator for intracerebral changes within patients with acute or chronical liver failure and before cerebral edema is developed in HE.

Moreover, it is also asserted that S100β increase in serum concentration can foresee HE. Additionally, there are limited evidences to prove S100β levels and existence of HE.

NSE is an CNS protein which exists in neurons and neuroendocrine tissues. NSE plays a role in glycolytic route in neurons as intracytoplasmic enzyme increasing serum level in case of neuron damage. Whilst S100β is the marker of astroglia dysfunction, NSE is the marker of neuronal dysfunction.

The aim of the study is analyzing S100β serum concentrations and correlate neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplantation candidates shall be accepted into the study.

Exclusion Criteria:

* Patients who:

Refused the study With infection, oncological and hematological diseases, coronary or kidney failure, malnutrition or skull fracture The ones who were transplanted liver from cadaveric Using psychoactive medicine Having respiratory system or central nerve system disease shall be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All living-made approximately 60 transplants shall be accepted.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Analyze S100β serum concentrations | before induction
  Blood sample is taken in preoperative period before induction of anesthesia in the operating room to analyze S100β serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.
Analyze S100β serum concentrations | first month
  Blood sample is taken first month in postoperative period to analyze S100β serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis
Analyze S100β serum concentrations | sixth month
  Blood sample is taken sixth month in postoperative period to analyze S100β serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.

SECONDARY OUTCOMES:
Analyze Neuron specific Enolase serum concentrations | before induction
  Blood sample is taken in preoperative period before induction of anesthesia in the operating room to analyze Neuron specific Enolase serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.
Analyze Neuron specific Enolase serum concentrations | first month
  Blood sample is taken first month in postoperative period to analyze Neuron specific Enolase serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.
Analyze Neuron specific Enolase serum concentrations | sixth month
  Blood sample is taken sixth month in postoperative period to analyze Neuron specific Enolase serum concentrations and neurologic damage of liver transplantation patients besides evaluating its effect on prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Medical Faculty Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The aim of the study is to evaluate neurological damage and analyze its effect on prognosis by considering S100β and NSE levels in liver transplantation.